CLINICAL TRIAL: NCT01862900
Title: Phase I/II Study of Stereotactic Body Radiation Therapy to Metastatic Lesions in the Liver or Lung in Combination With Monoclonal Antibody to OX40 (MEDI6469) in Patients With Progressive Metastatic Breast Cancer After Systemic Therapy.
Brief Title: Stereotactic Body Radiation and Monoclonal Antibody to OX40 (MEDI6469) in Breast Cancer Patients With Metastatic Lesions
Acronym: OX40 Breast
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: Robert W. Franz Cancer Center (Unknown); Providence Cancer Center, Earle A. Chiles Research Institute (Other); MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-017A; NCT01642290 (obsolete NCT alias)
Record Dates: First submitted 2013-05-22; First posted 2013-05-27 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2018-08

CONDITIONS: Metastatic Breast Cancer; Lung Metastases; Liver Metastases
Keywords: Breast Cancer; Metastatic; Lung metastases; Liver metastases; Stereotactic body radiation; anti-OX40 antibody; MEDI6469; Immunotherapy
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 15 Gy (Experimental): Patients receive a radiation dose of 15 Gy to their liver or lung metastases. Patients receive a dose of MEDI6469 following radiation and on Days 3, and 5.
  Interventions: Biological: MEDI6469
- 20 Gy (Experimental): Patients receive a radiation dose of 20 Gy to their liver or lung metastases. Patients receive a dose of MEDI6469 following radiation and on Days 3, and 5.
  Interventions: Biological: MEDI6469
- 25 Gy (Experimental): Patients receive a radiation dose of 25 Gy to their liver or lung metastases. Patients receive a dose of MEDI6469 following radiation and on Days 3, and 5.
  Interventions: Biological: MEDI6469

INTERVENTIONS:
Biological: MEDI6469 — Patients receive 3 doses of MEDI6469; one on Days 1, 3, and 5

SUMMARY:
This study will test the investigational antibody, MEDI6469 (anti-OX40), in combination with stereotactic body radiation in breast cancer patients that have liver or lung metastases and have received systemic therapy and have progressive disease. The investigators hypothesize that SBRT directed at metastatic breast cancer lesions will result in a systemic anti-tumor immune system response. This amplified and directed immune response could result in anti-tumor responses.

DETAILED DESCRIPTION:
Patients will receive one of three different doses of SBRT depending on which cohort they are in. The doses are:

Cohort 1: 15 Gy (central tumors 10 Gy); Cohort 2: 20 Gy (central tumors 15 Gy); Cohort 3: 20 Gy x 2 (central tumors 15 Gy x 2).

In addition, all patients will receive three doses of MEDI6469. MEDI6469 is administered at 0.4 mg/kg IV over 60 minutes using in-line filter on Days 1, 3, and 5.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast cancer with clinical evidence of stage 4 disease
* Measurable disease and at least one lesion in either liver or lung that is amenable to stereotactic body radiation
* One site of disease that will not receive radiation
* Patients with hormone receptor positive breast cancer must have received prior anti-hormonal therapy for metastatic disease and have progressed and patients with hormone receptor negative breast cancer must have received at least one prior chemotherapy regimen and progressed.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
* Women of childbearing potential must have a negative pregnancy test on the day treatment starts and must avoid becoming pregnant while on treatment. Men must avoid fathering a child while on treatment.
* Patients must have blood test results within pre-specified range
* No active bleeding
* No clinical coagulopathy (INR <1.5, PT <16 seconds, PTT < 38 seconds) within 28 days
* Anticipated lifespan greater than 12 weeks

Exclusion Criteria:

* Active infection requiring systemic antibiotics.
* Active autoimmune disease as defined by the autoimmune disease assessment tool.
* Previous treatment with mouse monoclonal antibodies
* At least 28 days since prior chemotherapy or monoclonal antibody therapy (trastuzumab or bevacizumab). Patients who have been on hormonal therapy can continue on therapy at the discretion of the investigator. Bisphosphonate therapy is acceptable during study participation.
* Diagnosis of a solid tumor malignancy (excluding non-melanoma skin cancer) within 3 years of enrollment.
* Need for chronic maintenance oral steroids.
* Active brain metastatic disease. Treated brain metastases with surgery, gamma-knife radiosurgery or radiation and stable for at least 4 weeks and off steroids are eligible.
* No metastatic site amenable to SBRT
* Pregnant or lactating women, as treatment involves risks to the embryo or fetus.
* Other medical or psychiatric conditions that in the opinion of the Principal Investigator would preclude safe participation in protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-04-27 (Actual); Primary Completion 2016-05-17 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose and safety profile of radiation administered in combination with anti-OX40 in patients with metastatic breast cancer. | From Day 1 to Day 36
  A dose limiting toxicity (DLT) is defined as any greater than or equal to grade 3 non-hematologic toxicity (except hypothyroidism or vitiligo) that in the opinion of the investigator is considered at least possibly related to treatment. Grade 3 or 4 hematologic toxicities that take longer than 10 days to resolve will be considered DLTs. Patients will have 8 clinic visits over 36 days to identify toxicities.

SECONDARY OUTCOMES:
Estimate the response rate of combined modality treatment in both irradiated and non-irradiated tumors. | Day 36
  Patients will have CT scans for tumor measurements at Day 36. Patients achieving a radiographic response, or are stable, will be followed monthly with physical exam and laboratory studies with CT (or other imaging as deemed appropriate) scans obtained every 3 months (± 2 weeks) for up to 24 months and then ever 6 months (± 2 weeks) for up to 4 years.

OTHER OUTCOMES:
Determine the influence of anti-OX40 and radiation on circulating CD4+ and CD8+ T cells. | Screening to Day 36
  Patients will provide 9 blood samples over 36 days to measure the number of CD4+ and CD8+ T Cells.

CONTACTS AND LOCATIONS:
Overall Officials: Marka R Crittenden, MD, PhD, Principal Investigator — Providence Cancer Center, Earle A. Chiles Research Institute; Brendan Curti, MD, Principal Investigator — Providence Cancer Center, Earle A. Chiles Research Institute; Steven Seung, MD, Principal Investigator — Providence Cancer Center, Earle A. Chiles Research Institute; Alison Conlin, MD, Principal Investigator — Providence Cancer Center, Earle A. Chiles Research Institute
Locations (1):
- Portland Providence Medical Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Providence Cancer Center — http://oregon.providence.org/patients/programs/providence-cancer-center-clinical-trials/Pages/default.aspx